CLINICAL TRIAL: NCT00123955
Title: Exercise Intolerance in Elderly Diastolic Heart Failure
Brief Title: PIE II: Pharmacological Intervention in the Elderly II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG0030; R01AG018915 (NIH); 2R01AG018915-05 (NIH)
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Diastolic Heart Failure; Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Spironolactone
  Interventions: Drug: Spironolactone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — 25mg tablet daily for 9 months
  Other Names: Aldactone
  Arms: 1
Drug: Placebo — Placebo tablet daily for 9 months
  Arms: 2

SUMMARY:
The purpose of this study is to examine whether spironolactone will improve exercise tolerance and quality of life in elderly patients with heart failure preserved ejection fraction (HFPEF).

DETAILED DESCRIPTION:
Exercise intolerance due to HFPEF is a major cause of disability among older Americans. Several lines of evidence suggest that aldosterone antagonism may improve exercise tolerance in HFPEF. Therefore, the primary aim of this study is to test the hypothesis that spironolactone will improve exercise tolerance and quality of life in elderly patients with isolated HFPEF. A total of 72 participants aged 60 or older will be randomized to receive either spironolactone 25mg daily or a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Medically stable
* Ages 60 or older
* Diagnosis of diastolic heart failure

Exclusion Criteria:

* Valvular heart disease
* Significant change in cardiac medication within the past 4 weeks
* Uncontrolled hypertension
* Recent or debilitating stroke
* Cancer or other noncardiovascular conditions with life expectancy less than 2 years
* Anemia
* Elevated serum potassium
* Renal insufficiency
* Psychiatric disease (uncontrolled major psychoses, depression, dementia, or personality disorder)
* Allergy to spironolactone; currently taking spironolactone or any aldosterone antagonist
* Plans to leave area within 1 year
* Refuses informed consent
* Failure to pass screening tests: pulmonary function, echocardiogram, or exercise
* Contra-indications to magnetic resonance imaging [MRI] (indwelling metal-containing prosthesis; pacemaker or defibrillator; history of welding occupation; uncontrollable claustrophobia)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-04; Primary Completion 2009-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W. Kitzman, MD, Principal Investigator — Professor of Internal Medicine, Cardiology, Director of Echocardiography, Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Kitzman DW, Little WC, Brubaker PH, Anderson RT, Hundley WG, Marburger CT, Brosnihan B, Morgan TM, Stewart KP. Pathophysiological characterization of isolated diastolic heart failure in comparison to systolic heart failure. JAMA. 2002 Nov 6;288(17):2144-50. doi: 10.1001/jama.288.17.2144. PMID 12413374
- [Background] Kitzman DW, Higginbotham MB, Cobb FR, Sheikh KH, Sullivan MJ. Exercise intolerance in patients with heart failure and preserved left ventricular systolic function: failure of the Frank-Starling mechanism. J Am Coll Cardiol. 1991 Apr;17(5):1065-72. doi: 10.1016/0735-1097(91)90832-t. PMID 2007704
- [Background] Kitzman DW, Gardin JM, Gottdiener JS, Arnold A, Boineau R, Aurigemma G, Marino EK, Lyles M, Cushman M, Enright PL; Cardiovascular Health Study Research Group. Importance of heart failure with preserved systolic function in patients > or = 65 years of age. CHS Research Group. Cardiovascular Health Study. Am J Cardiol. 2001 Feb 15;87(4):413-9. doi: 10.1016/s0002-9149(00)01393-x. PMID 11179524
- [Background] Zannad F, Alla F, Dousset B, Perez A, Pitt B. Limitation of excessive extracellular matrix turnover may contribute to survival benefit of spironolactone therapy in patients with congestive heart failure: insights from the randomized aldactone evaluation study (RALES). Rales Investigators. Circulation. 2000 Nov 28;102(22):2700-6. doi: 10.1161/01.cir.102.22.2700. PMID 11094035
- [Background] Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999 Sep 2;341(10):709-17. doi: 10.1056/NEJM199909023411001. PMID 10471456
- [Background] Cicoira M, Zanolla L, Franceschini L, Rossi A, Golia G, Zeni P, Caruso B, Zardini P. Relation of aldosterone "escape" despite angiotensin-converting enzyme inhibitor administration to impaired exercise capacity in chronic congestive heart failure secondary to ischemic or idiopathic dilated cardiomyopathy. Am J Cardiol. 2002 Feb 15;89(4):403-7. doi: 10.1016/s0002-9149(01)02261-5. PMID 11835920
- [Background] Kitzman DW, Herrington DM, Brubaker PH, Moore JB, Eggebeen J, Haykowsky MJ. Carotid arterial stiffness and its relationship to exercise intolerance in older patients with heart failure and preserved ejection fraction. Hypertension. 2013 Jan;61(1):112-9. doi: 10.1161/HYPERTENSIONAHA.111.00163. Epub 2012 Nov 12. PMID 23150511
- [Background] Daniel KR, Wells G, Stewart K, Moore B, Kitzman DW. Effect of aldosterone antagonism on exercise tolerance, Doppler diastolic function, and quality of life in older women with diastolic heart failure. Congest Heart Fail. 2009 Mar-Apr;15(2):68-74. doi: 10.1111/j.1751-7133.2009.00056.x. PMID 19379452

RESULTS

PARTICIPANT FLOW:
Groups:
- Spironolactone: Spironolactone
  Spironolactone: 25mg tablet daily for 9 months
- Placebo: Placebo
  Placebo: Placebo tablet daily for 9 months
Period: Overall Study
Arm/Group | Spironolactone | Placebo
Started | 42 | 38
Completed | 37 | 34
Not Completed | 5 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Placebo | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (7.3) | 71.7 (7.3) | 70.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 8 | 8 | 16
Peak VO2 (ml/kg/min) [Mean (Standard Deviation); unit: ml/kg/min] | 13.5 (2.9) | 13.3 (2.9) | 13.4 (2.9)
Workload (Watts) [Mean (Standard Deviation); unit: Watts] | 63 (26) | 60 (26) | 62 (26)

OUTCOME MEASURES:

1. Primary Outcome: Exercise Intolerance
Description: Peak exercise VO2
Time Frame: Baseline, 4 and 9 months
Population: The outcome measure data uses data from all participants with 4 and/or 9 month follow-up. Thirty-seven participants randomized to spironolactone and 35 participants randomized to placebo completed 4 months of follow-up, and 37 participants randomized to spironolactone and 34 participants randomized to placebo completed 9 months of follow-up.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 37 | 35
ml/kg/min
  Baseline | 13.5 (2.9) | 13.3 (2.9)
  4 months | 13.6 (3.5) | 13.5 (3.4)
  9 months: number analyzed (Participants) | 37 | 34
  9 months | 13.8 (3.2) | 13.9 (3.7)

2. Primary Outcome: Quality of Life Measured by the Minnesota Living With Heart Failure Questionnaire-total Score
Description: The Minnesota Living with Heart Failure Questionnaire (MLHF) is a self-administered disease-specific questionnaire for patients with Heart Failure, comprising 21 items rated on six-point Likert scales, representing different degrees of impact of HF on HRQoL, from 0 (none) to 5 (very much). It provides a total score (range 0-105, from best to worst HRQoL), as well as scores for two dimensions, physical (8 items, range 0-40) and emotional (5 items, range 0-25). The other eight items (of the total of 21) are only considered for the calculation of the total score.
  Scale of 0-105:The higher the score the worse the heart failure related Quality of Life.
Time Frame: Baseline, 4 and 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 37 | 35
units on a scale
  Baseline | 32 (21) | 28 (19)
  4 months | 29 (20) | 29 (23)
  Final- 9 months | 29 (18) | 25 (18)

3. Secondary Outcome: Concentric Left Ventricular Remodeling
Description: Left ventricle measurements by MRI:
  Mass/end diastolic volume ratio: g/ml
Time Frame: Baseline, 9 month
Measure: Mean (Standard Deviation); unit: g/ml
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 37 | 35
g/ml
  baseline | 1.8 (.4) | 1.7 (.5)
  9 month | 1.7 (.4) | 1.6 (.4)

4. Secondary Outcome: Left Ventricular Diastolic Stiffness
Description: Echocardiography Doppler measurement of left ventricular diastolic function:
  Early mitral annulus velocity (lateral) (Ea; cm/s)
Time Frame: Baseline, 4 month and 9 month
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 37 | 35
cm/s
  baseline | 7.0 (2.1) | 6.8 (1.4)
  4 month | 7.0 (2.1) | 6.8 (1.4)
  9 month | 7.4 (2.2) | 6.6 (1.6)

ADVERSE EVENTS:
Arm/Group | Spironolactone | Placebo
Serious Adverse Events (participants affected / at risk) | 6/42 | 6/38
Other Adverse Events (participants affected / at risk) | 0/42 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spironolactone (N=42) | Placebo (N=38)
Hospitalization for chest pain (Cardiac disorders) | 2 (2) | 1 (1)
Elective surgery (General disorders) | 1 (1) | 3 (3)
Hospitalization for shortness of breath (Cardiac disorders) | 0 (0) | 3 (5)
Hospitalization for syncope (Cardiac disorders) | 2 (2) | 0 (0)
Hospitalization for hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization for angioedema (Vascular disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) — Motor vehicle accident

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes